CLINICAL TRIAL: NCT06340659
Title: Concurrent Aerobic Exercise and Cognitive Training to Prevent Alzheimer's in At-risk Older Adults (The Exergames Telerehabilitation Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: AE and CT
Record Dates: First submitted 2024-03-08; First posted 2024-04-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: At Risk for AD-dementia, With Subjective Cognitive Decline

STUDY DESIGN:
Intervention Model Description: This study will use a single-blind, randomized trial will randomize 104 community-dwelling older adults to one of two arms for 3 months: home-based (asynchronous) Exergame (HbExergame) or home-based asynchronous aerobic exercise (HbAEx). Randomization will allocate subjects on a 1:1 allocation ratio within each age stratum (65-74 and ≥75) in random blocks of 8 or 4
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Subjects randomized to HbAEX
  Interventions: Behavioral: HbAEx
- Group 2 (Experimental): Subjects randomized to HbExergame
  Interventions: Behavioral: HbExergame

INTERVENTIONS:
Behavioral: HbAEx — Participants will have a 1-week (3 session) on-boarding period where study interventionists will deliver all necessary equipment (bike, pulse oximeters, etc.) to the participants' home, review the AEx program and prescription, and supervise the first 3 sessions to ensure participant understanding and fidelity of the AEx program. Thereafter, the remaining 33 sessions will be conducted by the participant without the direct supervision (asynchronous telerehabilitation) of the study interventionists. Subjects will cycle on recumbent stationary cycles at moderate-vigorous intensity individualized as 50-70% of heart rate reserve (HRR) and/or 11-14 on Borg Category Ratio-15 Rating of Perceived Exertion (RPE) Scale, for 30-50 minutes per session. Following the completion of each session, during the check-in meeting with the participant, the study interventionist will gather information from the participant (including HR and RPE) for dose quantification.
  Arms: Group 1
Behavioral: HbExergame — Participants will cycle as described in the HbAEx protocol while engaging in cognitive training for the duration of cycling. Cognitive training will include 20 levels of difficulty with 8-10 task scenarios in the context of three virtual worlds (environments. In each of the environments, the participant must follow directions and navigate to a destination where the scenario (cognitive task) will be performed. The game will inform the participant of the assigned task and, automatically, determine and inform the participant of the fastest route from the starting point to the scenario destination where the task will be performed. The participant will be required to remember the assigned task, follow the directions and navigate to the destination, and then remember what action is required to complete the task. A scenario-specific cognitive task will be triggered once the destination has been reached. The cycling and cognitive tasks will be completed throughout the sessions.
  Arms: Group 2

SUMMARY:
Significance of Research Question/Purpose: Subjective cognitive decline (SCD) is regarded as the first clinical manifestation in the AD-dementia continuum and currently has a prevalence of 11.2% in adults over the age of 45, with incidence increasing with greater age. Furthermore, population-based studies suggest that between 50% and 80% of older individuals (aged 70 years and older) who perform normally on cognitive tests, report some form of perceived decline in cognitive functioning when asked. The SCD state is unique as this population is more likely than their healthy peers to present with AD biomarkers such as neurodegeneration and amyloid burden, and therefore represents probable preclinical AD relative to other causes of SCD. Likewise, growing evidence suggests that a significant proportion of those adults are subsequently found to develop MCI, or AD, following the classic SCD-MCI-AD trajectory, with SCD increasing MCI risk 1.5-3 fold. Preventing Alzheimer's disease (AD) is arguably the most important approach to address the dementia epidemic worldwide because 99.6% of drug trials failed and no drugs can yet prevent, cure, or even slow AD. A treatment that delays the onset of AD by five years could save $89 billion in 2030.This highlights an urgent and pressing need to develop behavioral interventions to prevent AD and slow its progression.

This study will use a randomized, 2-parallel group, trial design that is guided by the Consolidated Standards of Reporting Trials (CONSORT)and the SPIRIT checklist. We will randomize 104 community-dwelling older adults to one of two arms for 3 months: home-based (asynchronous telerehabilitation) Exergame (HbExergame) or home-based (asynchronous telerehabilitation) aerobic exercise (HbAEx). Randomization will allocate subjects on a 1:1 allocation ratio within each age stratum (65-74 and >75), and will use permuted blocks of 8 and 4. We do not expect equal numbers of subjects in each age stratum, but want to balance the groups for each age. Investigators will be blinded to group assignment. All participants will be blinded to study aims and reminded as needed not to discuss their experiences with outcome assessors. Outcome assessors (also blinded to group allocations) will measure: 1) feasibility (attendance, adherence to exercise dose, systems usability scale), 2) preliminary cognition: fluid cognition [primary outcome], attention, episodic memory, and processing speed [secondary outcomes] using the NIH Toolbox cognition battery and aerobic fitness [VO2peak and 6-minute walk distance], and 3) blood neurotrophic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive complaint (defined as answering yes to the questions's "Do you perceive memory or cognitve difficulties?" and "In the last two years, has your cognition or memory declined?";
* Montreal Cognitive Assessement (MoCA) 26 or greater
* Age 65 years and older;
* English-speaking;
* Without ACSM contraindication to exercise

Exclusion Criteria:

* Dementia or mild cognitive impairment diagnosis;
* Neurological or major psychiatric disorder, alcohol/chemical dependency or recent medical condition (anethesia COVID-19 ["brain fog"]) likely causing cognitive impairment;
* Current enrollment in another intervention study

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
fluid cognition (global cognition) | 12 weeks
  which refers to the overall cognitive ability and will be assessed with the NIH Toolbox Cognitive Battery (NIHTB-CB) and its Fluid Composite Score (convergent validity [r = 0.78] and test-retest reliability [r = 0.86)

SECONDARY OUTCOMES:
Aerobic fitness | 12 weeks
  Aerobic fitness will be evaluated by the shuttle walk test (SWT) and followed guidelines as described by Singh and colleagues. Assistive devices will be permitted, such as ankle braces, walkers, crutches, or canes. Participants will be instructed to walk a distance of 10 meters around a marking between two cones, placed 0.5 m from each endpoint.
Neuroprotective biomarkers and ApoE status. | 12 weeks
  Blood samples will be obtained by venipuncture from the antecubital vein. perform biochemical analyses of the following biomarkers: 1) peripheral neuroprotective biomarkers serum brain-derived neurotrophic factor (BDNF) and plasma IGF-1; (neurotrophic) IL-6 (systemic inflammation); glial fibrillary acidic protein (GFAP) (neuroinflammation) and, 2) APOE genotypes at the end of the study to minimize the overall variance in biochemical analyses.
Exergame-specific usability and satisfaction | 12 weeks
  For individuals randomized to the HbExergame groups, usability and satisfaction of the Exergame will be assessed via questionnaire.
  The Systems Usability Survey contains 14 usability- related questions using Likert scale format from 1-5 with verbal anchors of strongly disagree (1), somewhat disagree (2), neutral (3), somewhat agree (4), and strongly agree (5); 4 items are reverse scored. In addition the questionnaire contains 5 satisfaction-related questions using similar scale. Verbal anchors include: very unsatisfied (1), somewhat unsatisfied (2), neutral (3), somewhat satisfied (4), and very satisfied (5). Composite scores for usability and satisfaction will be quantified. A second questionnaire, The User Engagement Scale (Long Form) will be used to assess a quality of user experience characterized by the depth of a participant's cognitive, temporal, affective and behavioral investment when interacting with a digital system. The User Engagement Scale has 3
SCD Symptoms | 12 weeks
  The Subjective Cognitive Decline Questionnaire (SCD-Q), a 27-item questionnaire, assesses both subject and informant self-perceived subjective decline in memory, language, and executive function in the last two years.
Anxiety Symptoms | 12 weeks
  Anxiety symptoms will be measured with the Geriatric Anxiety Scale (GAS-10) a 10-item version Likert scale (0-3 with 3 representing increased symptoms). The total GAS-10 scores range from 0 (no anxiety) to 30 (severe anxiety). It is a reliable and valid assessment for assessing anxiety symptoms with overall adequate internal consistency (Cronbach's alpha of 0.93)
Depressive Symptoms | 12 weeks
  Depression symptoms will assessed with the 15-item dichotomous (yes/no) Geriatric Depression Scale Short Form (GDS-SF). The GDS-SF scores range from 0 (no depression) to 15 (severe depression). It is a reliable and valid assessment for assessing depression symptoms with overall adequate internal consistency (Cronbach's alphas of 0.74-0.76) and statistically significant construct validity (dimensionality coefficients of 0.94).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States